CLINICAL TRIAL: NCT02944838
Title: Senior Change Makers Study: Improving Physical Activity Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dilip V. Jeste, Distinguished Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 160954
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Sedentary Lifestyle
Keywords: older adults; physical activity; built environment
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advocacy (Active Comparator): The Senior Change Makers Advocacy Program consists of weekly meetings, 1 hour each, for 8-weeks. The program will be led by graduate level students and will address topics such as how the environment affects walking, potential pedestrian hazards and solutions, how to conduct an audit of the walking environment, what advocates do, local examples of successful advocacy projects, creating an advocacy action plan, creating a fact sheet about the advocacy issue, writing letters to representatives, and making an advocacy presentation. The program will culminate with the presentation of the advocacy issue to a "decision maker" (e.g., a city planner, engineer, city council member, etc.).
  Interventions: Behavioral: Senior Change Makers Advocacy Program
- Physical Activity (Active Comparator): The Senior Change Makers Physical Activity Program consists of weekly meetings, 1 hour each, for 8 weeks. The program provides participants with information about safe physical activity, strategies to increase physical activity, and guided walks. Topics will focus on walking, but we will also include information and activities relating to strength training, flexibility, and balance. Behavioral skills such as goal setting, addressing barriers, and social support will also be addressed.
  Interventions: Behavioral: Senior Change Makers Physical Activity Program

INTERVENTIONS:
Behavioral: Senior Change Makers Advocacy Program — see description
  Arms: Advocacy
Behavioral: Senior Change Makers Physical Activity Program — see description
  Arms: Physical Activity

SUMMARY:
Senior Change Makers is an intergenerational intervention that compares two, 8-week programs: (1) an advocacy program wherein senior participants perform audits of their physical activity environments, identify an advocacy project, and advocate for improvements; and (2) a walking program designed to increase participant physical activity through education and guided walks. The investigators expect that the advocacy program will produce greater improvements in seniors' advocacy skills, confidence, and attitudes at 8 weeks.

DETAILED DESCRIPTION:
The proposed study will be conducted at six senior centers in San Diego, California and will involve 132 senior participants, 16 student participants, and 12 decision maker participants (N = 160). Three senior centers will be randomized to an advocacy program and three will be randomized to a walking program.

The participants at the advocacy intervention sites will undergo an 8-week advocacy program during which they will (1) learn about the connection between the built environment and physical activity, (2) conduct a field audit of their physical activity environment using the Microscale Audit of Pedestrian Streetscapes (MAPS) Mini tool, (3) select an advocacy issue related to a physical activity barrier, and (4) engage in advocacy actions, such as communicating with decision makers or public officials. The group sessions will include topics such as how the environment affects walking, potential pedestrian hazards and solutions, how to conduct an audit of the walking environment, what advocates do, local examples of successful advocacy projects, creating an advocacy action plan, creating a fact sheet about the advocacy issue, writing letters to representatives, making an advocacy presentation. The student participants will work with the senior participants throughout the program to help accomplish the advocacy goals. The program will culminate with the presentation of the advocacy issue to a "decision maker" (e.g., a city planner, engineer, city council member, etc.).

In the other study condition, the walking groups, participants will undergo an 8-week program that provides participants with information about safe physical activity, strategies to increase physical activity, and guided walks. The group sessions will address topics such as the benefits of walking, fall prevention tips, goal setting, positive thinking, social support, sedentary behavior and health, barriers to walking, handling setbacks, and overcoming challenges to physical activity. Comparing two beneficial programs helps with participant recruitment and retention, and ensures that between-group differences in outcomes are not due solely to participation in a group program.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* have not had a fall that resulted in a hospitalization in the past 12 months
* able to walk 3 meters within 30 seconds (Shumway-Cook, et al., 2000)
* able to walk without human assistance (cane or walker use okay)
* able to read and write in English
* able to complete written surveys without assistance
* able to attend regular study activities at the center
* able to provide written informed consent

Exclusion Criteria:

* Older adult participants will be excluded if they:
* are younger than 50 years
* have had a fall that resulted in a hospitalization in the last 12 months
* cannot complete the walking test within 30 seconds
* are not able to read and write in English
* are not able to complete written surveys without assistance
* cannot regularly attend study activities at the center
* are not willing to complete study activities
* are not willing to complete study assessment and wear the activity meter
* are not able to provide written informed consent
* cannot walk without human assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Advocacy skills and beliefs | 8 weeks
  The investigators will use validated survey items to measure seniors' changes in self-efficacy for advocacy, perceived socio-political control, and assertiveness (Millstein, 2013). Sample item: "I am confident that I can work to make my community a better place for being physically active." These are key outcomes of the advocacy training

SECONDARY OUTCOMES:
Intergenerational attitudes | 8 weeks
  Senior and student participants will complete pre-post survey items to assess changes in intergenerational attitudes and beliefs.
Advocacy actions and outcomes | 8 weeks and 3 months
  The investigators will measure completion of advocacy "actions" and "outcomes" with a checklist survey taken by the researchers. Examples of actions include testimony, letters, and meetings. To determine if decision makers took any action after the advocacy, the investigators will ask the decision makers or their staff to complete a short, 10-minute survey, after the advocacy action. The survey will solicit feedback for the advocates, assess whether any action occurred, and assess the decision makers' perceptions of the advocacy and study. Researchers will follow-up again at 3 months to assess completion of advocacy actions, if the decision makers took any actions, and whether any changes occurred
Physical activity | 8 weeks
  Physical activity will be measured at baseline and after completion of the 8-week intervention. The investigators will use Actigraph accelerometers (model GT3X, Pensacola, FL), set to collect data in 60 second epochs to match cut points. Senior participants will wear the accelerometer for seven days during all waking hours (except when bathing or swimming) and estimates of physical activity levels and sedentary time will be calculated using validated algorithms and cut points for seniors.

CONTACTS AND LOCATIONS:
Overall Officials: James Sallis, PhD, Principal Investigator — Distinguished Professor; Dilip Jeste, PhD, Principal Investigator — Distinguished Professor
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patch CM, Conway TL, Kerr J, Arredondo EM, Levy S, Spoon C, Butte KJ, Sannidhi D, Millstein RA, Glorioso D, Jeste DV, Sallis JF. Engaging older adults as advocates for age-friendly, walkable communities: The Senior Change Makers Pilot Study. Transl Behav Med. 2021 Sep 15;11(9):1751-1763. doi: 10.1093/tbm/ibab098. PMID 34293156